CLINICAL TRIAL: NCT03544164
Title: Assessing Respiratory Rate and Tidal Volume Delivery During Manual Ventilation
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Brady Scott, Assistant Professor, Director of Clinical Education, Rush University Medical Center
Other Study IDs: 18020603
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Advanced Cardiac Life Support, Cardiopulmonary Resuscitation, Tidal Volume, Manual Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Manual Ventilation — Manual ventilation via endotracheal tube using adult manual resuscitation device

SUMMARY:
Excessive minute ventilation for patients who experience cardiac arrest may cause pulmonary injury and decrease the overall effectiveness of cardiopulmonary resuscitation (CPR). Although clinicians are trained with the correct technique for manual ventilation, evidence still shows that clinicians tend to deliver a higher respiratory rate than recommended during CPR. Little is known about tidal volume delivery during CPR; either the amount of volume give or even the impact of tidal volume on the effectiveness of CPR. There are many factors that may influence variations of tidal volumes and RR during CPR. These factors include distractions in the room (noise/cross talk), inability to assess tidal volume delivery, anxiety, and stress of the situation. This study will evaluate tidal volume and respiratory rate (RR) delivery during a simulated CPR situation. Participants will be asked to provide care for an intubated adult patient in cardiac arrest, which will include all components of advanced cardiac life support training.

DETAILED DESCRIPTION:
This will be a cross-sectional study, conducted during regularly scheduled ACLS courses at Rush University Medical Center. Enrollment will be by random assignment as participants arrive for the ACLS course. Those that consent to the study will be informed that the investigator's study is to observe ACLS performance, but the exact parameters being measured will not be disclosed in an effort to mitigate any changes in behaviors.

During the course of the study, groups will be assigned sequentially, and the first group to participate will be termed as "Group 1". Within the group, each participant will be assigned a letter to identify the sequence of rotation with the skills. For example, the first participant in group 1 to perform manual ventilation will be assigned the study identity of "1A". The second person in the first group will be "1B", and so on.

During the ACLS megacode component of the ACLS training, each study participant will be given the opportunity to manually ventilate the simulated intubated adult patient, as per the normal rotation during a megacode. During the megacode, information will be collected via the NICO2 Respiratory Management System (Philips Respironics, Murrysville, Pennsylvania) that is attached to the endotracheal tube, which will be video recorded, as this system does not have function of data storage or downloaded. This is to assure each breath is captured so the study team can assure accuracy of data collection. None of the study participants will be video recorded.

At the completion of the study, each participant will be debriefed on their performance and informed of the true nature of the study; which is to evaluate respiratory rate and tidal volume delivery during manual ventilation to an intubated patient during an ACLS rescue attempt.

ELIGIBILITY:
Inclusion Criteria:

* 21 years old or older
* licensed clinician, regardless of medical profession

Exclusion Criteria:

* Full-time, non-licensed students that have no completed their formal training program at Rush University

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical professionals attending an American Heart Association Advanced Cardiac Life Support course
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-07-07 (Actual); Study Completion 2019-07-07 (Actual)

PRIMARY OUTCOMES:
Tidal Volume delivery | through study completion, an average of 1 year
  Amount of volume delivered in milliliters per squeeze of the resuscitation device

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No